CLINICAL TRIAL: NCT07388121
Title: The Effect of Vitamin C Supplementation on Gut Microbiota Composition and Metabolic Activity in Healthy Adults
Brief Title: The Effect of Vitamin C Supplementation on Gut Microbiota Composition and Function in Healthy Adults
Acronym: VitaGut
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Glasgow (Other)
Collaborators: Professor Konstantinos Gerasimidis, University of Glasgow (Unknown)
Responsible Party: Principal Investigator, Athanasios Koutsos, Lecturer in Human Nutrition, University of Glasgow
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 200250024
Record Dates: First submitted 2025-12-18; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-11

CONDITIONS: Short Chain Fatty Acids Concentration in Stools; Gut Microbiota Diversity and Composition
Keywords: vitamin C; gut microbiota; SCFA
MeSH Terms: interventions — Jogging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sequential vitamin C intervention (Experimental): In this single-arm, sequential dietary intervention study, participants will follow their normal habitual diet for one week (run-in period) and then receive two different doses of vitamin C tablets over two consecutive 14-day periods: a moderate dose of 200 mg/day during the first period (2 weeks) and a high dose of 1000 mg/day during the second period (another 2 weeks). The study also includes one week post intervention follow up period (habitual diet) after the high vitamin C dose where participants return to their habitual diet without vitamin C supplementation
  Interventions: Dietary Supplement: Moderate Vitamin C dose (200 mg); Dietary Supplement: High-dose vitamin C supplementation (1000 mg); Other: Habitual diet (run in period)

INTERVENTIONS:
Dietary Supplement: Moderate Vitamin C dose (200 mg) — 200 mg of vitamin C provided as a chewable tablet, taken orally daily for two weeks
Dietary Supplement: High-dose vitamin C supplementation (1000 mg) — 1000 mg of Vitamin C provided as a chewable tablet, taken orally daily for two weeks
Other: Habitual diet (run in period) — this is a run-in period where participants consume their habitual diet for one week

SUMMARY:
The aim of this dietary intervention study is to explore how vitamin C affects the bacteria that live in our gut. Vitamins are essential nutrients found in fruits and vegetables. Our bodies cannot make them on their own, but we need them to function correctly. Vitamins play various roles, including supporting the immune system and assisting with energy production. Some vitamins in our diet can reach the large intestine, where they may be used by gut bacteria to promote their growth. In this study, we aim to investigate how our gut bacteria interact with vitamin C and how this interaction affects their growth and activity.

For this study, participants will follow their habitual diet for one-week (run-in period), followed by two consecutive two-week supplementation periods in which they will first take a moderate dose (200 mg/day) and then a high-dose (1000 mg/day) of vitamin C. A final one-week period follow up period will involve a return to their habitual diet. Faecal, blood and urine samples will be collected at the start and end of each supplementation period to explore changes in gut microbiota composition, activity and markers of inflammation.

DETAILED DESCRIPTION:
This is a sequential dietary intervention trial exploring the effects of two doses of vitamin C supplementation on gut microbiota: a moderate, diet-achievable dose of 200 mg/day, and a high dose of 1000 mg/day, each given for two weeks. Primary outcomes will be gut microbiota activity (SCFA production) and composition while secondary exploratory outcomes will include systemic inflammation and gut barrier integrity markers. We anticipate that this pilot study will provide valuable insights into the dose-response effects of vitamin C and help define optimal intakes for promoting gut health.

Twenty-three healthy adults will be recruited from the Glasgow area, with all study visits taking place at the New Lister Building, University of Glasgow. Each participant will attend four study visits over six weeks.

The intervention includes:

* One-week run-in period (habitual diet)
* Two weeks of moderate-dose vitamin C (Vitamin C Chewable Tablet 200 mg, one tablet per day)
* Two weeks of high-dose vitamin C (Vitamin C Chewable Tablet 1000 mg, one tablet per day)
* One-week follow-up (habitual diet)

There will be no washout period between the study periods and participants will be instructed to maintain their usual diet and lifestyle throughout the trial.

Hypothesis Vitamin C supplementation will increase stool SCFAs, particularly butyrate, and beneficially modulate gut microbiota composition, systemic inflammation and gut barrier integrity in healthy adults.

Study schedule and sample collection:

* Visit 1 (Week 0): Baseline anthropometric measurements will be taken (height, weight, body composition); stool and urine sample collection will be arranged. Participants will follow habitual diet for one week (run-in period).
* Visit 2 (Week 1): Anthropometric measurements; stool sample, and fasted blood and urine samples will be collected. The participants will begin a moderate-dose vitamin C supplementation (Vitamin C Chewable Tablet 200mg, one tablet per day) for two weeks (moderate-dose period), in addition to their usual diet.
* Visit 3 (Week 3): Anthropometric measurements; stool sample, and fasted blood and urine samples will be collected. The participants will switch to a high-dose vitamin C supplementation (Vitamin C Chewable Tablet 1000mg, one tablet per day) for two weeks (high-dose period), in addition to their usual diet.
* Visit 4 (Week 5): Anthropometrics; stool sample, and fasted blood and urine samples will be collected. Participants will resume their habitual diet for one week (follow-up period).
* Follow up (Week 6): Final stool sample collected.

Three-day food diaries, Gastrointestinal Symptoms Rating Scale (GSRS) diary, and compliance tick sheets will be completed during the run-in, moderate-dose, and high-dose periods.

Sample size The sample size is based on anticipated effects on stool butyrate, a key SCFA expected to be modified by the intervention. Based on literature and our group's previous results, recruiting 20 healthy participants would provide 80% power (P=0.05) to detect a mean change of 4 μmol/g in stool butyrate (SD: 4.5 μmol/g). Allowing for 15% drop-out, a total of 23 participants will ensure adequate power.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals aged 18-65 years with a BMI between 18.5-35 Kg/m2
* Self-reported good health with no chronic conditions requiring regular medical care
* Willing to provide blood, urine, and stool samples at multiple time points

Exclusion Criteria:

* Aged <18 or >65 years
* Smoking
* Chronic illness requiring regular medication or GP visits
* Current or recent medication affecting gut transit or digestion
* Major gastrointestinal surgery
* Pregnant or breastfeeding
* Regular use of pre/probiotics, vitamins, or minerals (unless willing to discontinue 2-4 weeks prior)
* Antibiotics in past 3 months
* Weight change >±2 kg in past month
* Participation in other research likely to interfere with this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Butyrate (Short Chain Fatty Acid) | Baseline (Visit 1), Week 1 (Visit 2), Week 3 (Visit 3), Week 5 (Visit 4) and Week 6 (Visit 5)
  Quantified in stool samples using Gas Chromatography
Short Chain Fatty Acids i.e. acetate, propionate, butyrate, total | Baseline (Visit 1), Week 1 (Visit 2), Week 3 (Visit 3), Week 5 (Visit 4) and Week 6 (Visit 5)
  Quantified in stool samples using Gas Chromatography
Stool microbiota composition analysis | Baseline (Visit 1), Week 1 (Visit 2), Week 3 (Visit 3), Week 5 (Visit 4) and Week 6 (Visit 5)
  16S rRNA gene amplicon sequencing from faecal DNA extracts

SECONDARY OUTCOMES:
Stool pH | Baseline (Visit 1), Week 1 (Visit 2), Week 3 (Visit 3), Week 5 (Visit 4) and Week 6 (Visit 5)
  pH meter
Vitamin C in plasma | Week 1 (Visit 2), Week 3 (Visit 3), and Week 5 (Visit 4)
  Using validated analytical techniques
Inflammatory markers | Week 1 (Visit 2), Week 3 (Visit 3), and Week 5 (Visit 4)
  Using Elisa or multiplex assays

OTHER OUTCOMES:
Gut barrier function markers | Week 1 (Visit 2), Week 3 (Visit 3), and Week 5 (Visit 4)
  Quantified in plasma using standard enzyme-linked immunosorbent assay.

CONTACTS AND LOCATIONS:
Overall Officials: Athanasios Koutsos, PhD, Principal Investigator — Human Nutrition, School of Medicine, College of Medical, Veterinary, and Life Sciences, University of Glasgow
Locations (1):
- New Lister Building, Glasgow Royal Infirmary, 10-16 Alexandra Parade, G31 2ER, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided